CLINICAL TRIAL: NCT04570982
Title: Compassionate Use of Remdesivir and Convalescent Plasma Therapy for Treatment of COVID-19 Infection in Nepal : A Prospective Observational Study (Amended Protocol)
Brief Title: Clinical Protocol for Convalescent Plasma and Remdesivir Therapy in Nepal
Acronym: CPT-R-Nepal
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dr. Pradip Gyanwali,MD (Other Government)
Collaborators: Ministry of Health and Population, Nepal (Other Government)
Responsible Party: Sponsor-Investigator, Dr. Pradip Gyanwali,MD, Chief-Executive, Nepal Health Research Council
Organization: Nepal Health Research Council (Other Government)
Other Study IDs: NHRC2020-001
Record Dates: First submitted 2020-07-24; First posted 2020-09-30 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: COVID-19
Keywords: Convalescent Plasma; Remdesivir
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Convalescent Plasma with SOC: All patients will receive CPT and SOC
  Interventions: Biological: Convalescent Plasma

INTERVENTIONS:
Biological: Convalescent Plasma — The objective of this protocol is to provide a coordinated approach for distribution and guidance for safe and effective administration of convalescent serum with antibodies against SAR CoV-2 for treatment of patients with COVID-19 infection who are most likely to benefit from this investigational treatment and monitor them.

SUMMARY:
The objective of this compassionate use study is to provide access and evaluate the outcome of Remdesivir and COVID-19 convalescent plasma use in patients with COVID-19. This protocol provides a coordinated approach for distribution and guidance for safe and effective administration of Remdesivir and convalescent plasma with antibodies against SARS CoV-2 for treatment of patients with COVID-19 infection who are most likely to benefit from this investigational treatment and monitor them for the following specific objectives and outcomes:

SPECIFIC OBJECTIVES

1. Provide access to convalescent plasma for hospitalized patients with severe COVID-19 infection (compassionate use, expanded access program)
2. Monitor safety of the therapy with convalescent plasma containing antibodies against SAR CoV-2 and Remdesivir for hospitalized patients with severe COVID-19 infection
3. Evaluate outcomes in patients who received convalescent COVID-19 plasma therapy alone, Remdesivir alone, and both agents.

Study Design: This study will be a prospective, observational clinical study with an intention-to-treat, cross-over design. Comparison groups will be patients who received convalescent plasma vs. those who received Remdesivir. In addition, cross-over to convalescent plasma arm will be allowed for patients who continued to get worse even after receiving Remdesivir for more than 48 hours.

DETAILED DESCRIPTION:
ENROLLMENT Patients will be recruited from all COVID-19 treating hospitals of Nepal which are participating in this clinical study. All hospitalized patients with moderate to severe COVID-19 infection will be screened for Remdesivir Treatment and those with severe to life threatening COVID-19 infection will be screened for Convalescent plasma therapy.

Donors Convalescent plasma donors will be recruited from the record of the hospitals from where they were discharged. The COVID hospitals will be asked to collect names of recovered patients who have voluntarily shown interest to donate plasma. When possible donated plasma will be stored in respective hospitals or blood bank.

ELIGIBILITY:
A. INCLUSION CRITERIA

All patients:

1. Minimum 18 years of age
2. Laboratory-confirmed diagnosis of COVID-19 infection with PCR test positive for SARS-CoV-2
3. Hospitalized patients admitted to an acute care facility for the treatment of COVID-19
4. Signed informed consent provided by the patient or patient's healthcare proxy

   For Remdesivir:
5. Moderate to severe COVID-19 infection who require to be on oxygen supplementation

   For convalescent plasma therapy:

   A patient has to meet one of the following criteria to be eligible for receiving convalescent plasma therapy:
6. Severe or life-threatening COVID-19 infection, or judged by the treating provider to be at high risk of progression to severe or life-threatening disease
7. Patients who progress to severe or life threatening infection despite being on remdesivir for 48 hours or longer.

B. EXCLUSION CRITERIA

1. Under 18 years of age
2. Not confirmed with PCR test for COVID-19 infection
3. Cases not meeting criteria for severe or life-threatening COVID-19 infection
4. Any patient with contraindications for receiving plasma transfusion will not receive plasma
5. Any patient with contraindications for receiving Remdesivir will not receive Remdesivir
6. Patient's declination to enroll in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from all COVID-19 treating hospitals of Nepal which are participating in this clinical study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-07-30 (Actual); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Availability of convalescent plasma | 12 Weeks
  * percentage of donors who donated plasma versus those who were eligible for donation
  * percentage of patient who received plasma vs. requests received
Amount of Plasma | 12 Weeks
  - amount of plasma administered per patient
Demographics of recipients | 12 Weeks
  - type of patients receiving plasma therapy : Age in Years, Sex: M/F,
Co-morbidity of recipient | 12 Weeks
  - recipient comorbidities: Smoking, Diabetes, Heart disease, Chronic lung disease, chronic liver disease, cancer, organ transplant, HIV infection, TB. HIV, HBV, HCV, Syphillis
Donor status | 12 Weeks
  * donor health status: HIV, HBV, HCV, Syphillis
  * Donor status: duration after recovery from COVID-19, plasma antibody titer against SARS CoV-2
Adverse events of convalescent COVID-19 plasma and Remdesivir Therapy | 12 Weeks
  * any expected and unexpected adverse events during or after treatment (upto 7 days)
  * any other complications related or unrelated to plasma transfusion and Remdesivir during hospital stay
Hospital and ICU length of stay | 12 Weeks
  - number of days of hospital stay and ICU stay
Disposition of patients including survival | 12 Weeks
  - condition at discharge: complete recovery, partial recovery with complications, death

CONTACTS AND LOCATIONS:
Overall Officials: Pradip Gyanwali, MD, Study Chair — Nepal Health Research Council; Meghnath Dhimal, PhD, Study Director — Nepal Health Research Council; Janak Koirala, MD, MPH, Principal Investigator — Nepal Health Research Council
Locations (6):
- Nepal (6):
  - Narayani Hospital, Birgunj
  - Seti Provincial Hospital, Dhangadi
  - BP Koirala Institute of Health Sciences (BPKIHS), Dharān
  - Sukraraj Tropical Disease Hospital, Kathmandu
  - TU Teaching Hospital, Kathmandu
  - Bheri Provincial Hospital, Nepalgunj

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koirala J, Gyanwali P, Gerzoff RB, Bhattarai S, Nepal B, Manandhar R, Jha R, Sharma S, Sharma YR, Bastola A, Murphy H, Acharya S, Adhikari P, Rajkarnikari M, Vaidya KM, Panthi CL, Bista B, Giri G, Aryal S, Pant S, Pokharel A, Karki S, Basnet S, Koirala B, Dhimal M; Nepal COVID-19 Clinical Study Collaborators. Experience of Treating COVID-19 With Remdesivir and Convalescent Plasma in a Resource-Limited Setting: A Prospective, Observational Study. Open Forum Infect Dis. 2021 Aug 21;8(8):ofab391. doi: 10.1093/ofid/ofab391. eCollection 2021 Aug. PMID 34430672